CLINICAL TRIAL: NCT00002003
Title: Phase II Study of Novantrone(R) (Mitoxantrone) and Etoposide in Patients With HIV Associated Large Cell and Immunoblastic Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lederle Laboratories (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 055A; 3-100
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-03

CONDITIONS: Lymphoma, Non-Hodgkin; HIV Infections
Keywords: Mitoxantrone; Lymphoma, Large-Cell; Etoposide; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; HIV Infections; Dendritic Cell Sarcoma, Interdigitating; Acquired Immunodeficiency Syndrome | interventions — Mitoxantrone; Etoposide

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride
Drug: Etoposide

SUMMARY:
To determine the efficacy and toxicity of the combination of mitoxantrone hydrochloride ( Novantrone ) and etoposide in the treatment of patients with HIV associated lymphomas.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Positive HIV antibody, positive HIV culture or antigen capture, or prior diagnosis of AIDS by the CDC criteria.
* Diagnosis by pathological examination of large cell or immunoblastic lymphoma within measurable or evaluable disease.
* Pneumocystis carinii pneumonia (PCP) prophylaxis during the course of the study.
* Signed written informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Acute intercurrent opportunistic infection, such as Pneumocystis carinii pneumonia (PCP) diagnosed within 3 weeks.
* Stage IE Central Nervous System lymphomas.

Patients with the following are excluded:

* More than one previous treatment for lymphoma.
* Acute intercurrent opportunistic infection, such as Pneumocystis carinii pneumonia (PCP) diagnosed within 3 weeks.
* Conditions that preclude obtaining an informed consent.
* Not accessible for scheduled treatment visits or follow-up.
* Stage IE Central Nervous System (CNS) lymphomas.

Prior Medication:

Excluded within 2 weeks of study entry:

* Zidovudine.
* Excluded:
* Doxorubicin dosing = or > 300 mg/m2.

Prior Treatment:

Excluded:

* Received more than one previous treatment regimen for lymphoma.

Required:

* Prophylactic treatment for Pneumocystis carinii pneumonia (PCP) prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UMDNJ - New Jersy Med School, Newark, New Jersey
  - New York Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York